CLINICAL TRIAL: NCT01397812
Title: Validation of Heartsbreath Test for Heart Transplant Rejection
Brief Title: Heartsbreath Test for Heart Transplant Rejection
Acronym: Heartsbreath
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Menssana Research, Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: MR-2011-03; 2R44HL059715-04A1 (NIH)
Record Dates: First submitted 2011-06-23; First posted 2011-07-20 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Heart Transplant Rejection
Keywords: Rejection of the Heart Transplant; Heart Transplant Rejection, an immune-mediated allograft injury; Non-cellular or humoral rejection in cardiac transplant recipients; Right ventricular endomyocardial biopsy to detect Heart transplant rejection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Subjects will comprise of patients who are the recipients of a heart transplant within the previous 12 months and are scheduled for a routine endomyocardial biopsy.
  Subjects will provide breath samples for the Heartsbreath test using the BreathScanner 1.0. Optionally subjects will provide breath samples using the BreathLink point of care system.
  Interventions: Device: BreathScanner 1.0; Device: BreathLink

INTERVENTIONS:
Device: BreathScanner 1.0 — For the HeartsBreath test, breath is collected using BreathScanner 1.0 and sent to central laboratory for analysis for markers of transplant rejection.
Device: BreathLink — The BreathLink point-of-care system detects and quantifies the breath VOC's determined to be biomarkers during the development of the Heartsbreath test.

SUMMARY:
The purpose of this study is to demonstrate and validate a breath test for detection of biomarkers of heart transplant rejection (Grade 2R heart transplant).

DETAILED DESCRIPTION:
This is a 36 month multi-center, open label, unblinded and blinded study on subjects have had a heart transplant within the previous 12 months and are scheduled to undergo an endomyocardial biopsy. The breath test will be performed to identify and validate the predicative algorithms that identify breath biomarkers for heart transplant rejection.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to cooperate with study, understand the scope of the study, and gives signed informed consent to participate.
* Subject is the recipient of a heart transplant within the previous 12 months
* Subject is scheduled for a routine endomyocardial biopsy
* Subject is 18 years or older

Exclusion Criteria:

* Evidence of acute intercurrent disease other than rejection reaction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject is the recipient of a heart transplant within the previous 12 months and is scheduled for a routine endomyocardial biopsy
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
To measure the sensitivity and specificity of the breath test as compared to the primary right ventricular endomyocardial biopsy for the development of an intrinsically safe, painless, and non-invasive detection technique. | 60 days after completion
  The current "gold standard" for heart transplant rejection diagnosis is a series of endomyocardial biopsies during the first twelve months after operation. This procedure is invasive, painful, and potentially hazardous. The Heartsbreath test is an intrinsically safe, painless, and non-invasive breath test for heart transplant rejection that employs volatile biomarkers of oxidative stress. The Food & Drug Administration (FDA) approved the Heartsbreath test for clinical use with a Humanitarian Device Exemption (HDE).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Phillips, MD, FACP, Principal Investigator — Menssana Research, Inc.
Locations (5):
- United States (5):
  - Cedars-Sinai Medical Center, Beverly Hills, California
  - Stanford University School of Medicine, Stanford, California
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Columbia Presbyterian Medical Center, New York, New York
  - Hahnemann University Hospital and the Drexel University College of Medicine, Philadelphia, Pennsylvania